CLINICAL TRIAL: NCT04512287
Title: A Randomized, Double-Blind, Placebo Controlled, Crossover Trial on Safety and Efficacy of Autologous Platelet-Rich Plasma for Treatment of Peyronie's Disease
Brief Title: PRP for Treatment of Peyronie's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Manuel Molina Leyba, Research Physician, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200779
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Peyronie Disease; Sexual Dysfunction, Physiological; Sexual Dysfunction Male; Genital Diseases, Male
Keywords: PD; PyD; PRP
MeSH Terms: conditions — Penile Induration; Sexual Dysfunction, Physiological; Genital Diseases, Male | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental: Autologous PRP followed by Placebo Group (Experimental): Participants in this group will receive the autologous intervention first, followed by the placebo intervention 3 months later.
  Interventions: Drug: Autologous Platelet Rich Plasma; Other: Saline Solution
- Experimental: Placebo followed by Autologous PRP Group (Experimental): Participants in this group will receive the placebo intervention first, followed by the Autologous PRP intervention 3 months later.
  Interventions: Drug: Autologous Platelet Rich Plasma; Other: Saline Solution

INTERVENTIONS:
Drug: Autologous Platelet Rich Plasma — 2 sessions of Autologous PRP will be administered 15 days apart. Each injection will be 0.5 mL of PRP injected into the Peyronie's disease penile plaque.
  Other Names: PRP
Other: Saline Solution — 2 sessions of saline injection will be administered 15 days apart. Each injection will be 0.5 mL of normal saline injected into the Peyronie's disease penile plaque.

SUMMARY:
The purpose of this study is to learn about the effects of Platelet-Rich Plasma (PRP) injection in men with Peyronie's Disease (PyD).

ELIGIBILITY:
Inclusion Criteria:

1. Be Male
2. Be 18 to 75 years of age (inclusive).
3. Be able to provide written informed consent
4. Have a diagnosis of PD with evidence of active or stable disease as determined by the investigator
5. Penile curvature deformity of >30° to <120°
6. Agree to comply with all study related tests/procedures.

Exclusion Criteria:

1. Previous penile surgery of any kind (except circumcision and condyloma removal), such as penile lengthening, penile cancer surgery, penile plication, grafting.
2. Previous intralesional injection therapy (such as Xiaflex) for PD.
3. Previous history of priapism or penile fracture
4. PD characterized by a ventral plaque
5. Severe erectile dysfunction as characterized with an International Index of Erectile Function (IIEF) score ≤ 16
6. Actively on anticoagulation during time frame of injections (aspirin 81 mg will be eligible for therapy)
7. Hour-glass deformity
8. Unwilling to participate
9. Medically unfit for sexual intercourse as deemed by the principal investigator
10. Patients scheduled to undergo an elective medical procedure during the investigation timeframe that will interfere with autologous PRP injection therapy.
11. Have a serious comorbid illness/condition/behavior that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects in each group who attain degree change in penile curvature. | 7 months
  Treatment efficacy of PRP will be assessed via the percentage of participants achieving degree change in penile curvature from baseline. Degree of curvature will be measured using a goniometer with the aid of injection of vasoactive substance into the penis.
Percentage of subjects achieving any decrease in PDQ sub-domain scores (Psychological and Physical Symptoms, Symptom Bother). | 7 months
  Treatment efficacy will be assessed via the percentage of participants achieving any decrease in Peyronie's disease Questionnaire (PDQ) sub-domain scoring from baseline. The sub-domains that will be assessed in primary outcome is Psychological and Physical Symptoms and Symptom Bother. PDQ is a validated 15-item questionnaire that assess Psychological and Physical Symptoms, Symptom Bother, and Penile Pain subdomains. The Psychological and Physical Symptoms subdomain is measured from 0 to 24 (most severe symptoms). Symptom Bother subdomain is measured from 0 to 30 (most severe pain).

SECONDARY OUTCOMES:
Incidence of adverse events in all patients | Baseline, 6 months (post-intervention)
  Safety will be evaluated via the incidence of adverse events as assessed by treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Molina, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chu KY, Molina ML, Ledesma B, Zucker I, Saltzman RG, Masterson TA, Ramasamy R. A Phase 2 Randomized, Placebo-controlled Crossover Trial to Evaluate Safety and Efficacy of Platelet-rich Plasma Injections for Peyronie's Disease: Clinical Trial Update. Eur Urol Focus. 2023 Jan;9(1):11-13. doi: 10.1016/j.euf.2022.08.017. Epub 2022 Sep 10. PMID 36100520